CLINICAL TRIAL: NCT03619720
Title: Production et Perception émotionnelle Chez Les Patients paralysés Faciaux: Marqueurs Respiratoires, Phonatoires et expressivité Faciale.
Brief Title: Emotional Perception and Production in Facial Palsy: Respiratory, Vocal and Facial Markers.
Acronym: ResPPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018-A01043-52
Record Dates: First submitted 2018-07-21; First posted 2018-08-08 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Facial Palsy
Keywords: Emotions, Respiratory Rate, Phonation
MeSH Terms: conditions — Facial Paralysis | interventions — Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental)
  Interventions: Other: Records

INTERVENTIONS:
Other: Records — Respiratory records, Vocal records Video records Questionnaires

SUMMARY:
Respiratory function, phonation and facial expressivity are related to emotional reaction through neurophysiological process. Specific emotional respiratory, vocal and facial patterns had been described in literature. Respiratory cycles variation is modulated by stimulus arousal. Furthermore, inspiratory-to-expiratory time ratio in abdominal area is modulated by emotional valence. Inextricably linked to respiration, vocal production depends on emotional arousal and valence too.

According to embodied cognition, the effector pattern of an emotion initiates the corresponding subjective activation. Facial recognition is influenced by automatic mimicry and facial feedback. Most facial feedback studies included patients with diplegia but few studies dealt with emotional perception in Bell's palsy.

The aim of the present study is to understand production and perception of emotion in Bell's palsy with respiratory, vocal and facial markers. What impact lack of mimicry have on physiological emotional reaction in Bell's palsy? To this end, prospective monocentric study will be conducted with 60 patients with Bell's Palsy from grade II to grade VI of House & Brackmann's scale. During production and perception of vocal and facial expression, respiratory rate and thoraco-abdominal movements will be analyzed. The investigators hypothesize that severity of facial deficit is negatively correlated with variation of respiratory cycles, lower segmental and suprasegmental changes during vocal expression, and lower facial perception (congruency and arousal).

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated to the health care system
* Patients must have been diagnosed with unilateral peripheral facial palsy stage III to VI, according to House and Brackmann international classification.
* To be able to read, understand and sign a consent
* To be able to understand French spoken and written

Exclusion Criteria:

* Diplegia or facial graft
* Visual disorders, non corrected
* Respiratory or vocal disorders
* Psychiatric history
* Facial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-11 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Effects of facial impairment on the respiratory rate | 1hour
  Facial impairment assesed with Sunnybrook Facial Grading Scale Composite Score in %.
  Respiratory rate is measured with chest and abdominal belt (breaths per minute).

SECONDARY OUTCOMES:
Effects of facial impairment on pitch variation (Hz) during emotional vocal production. | 1hour
  Acoustic measures lead with Praat Analysis software. Variation pitch between first and last segment of the emotional sentence calculated in Herz.
Effects of facial impairment on perception of emotional facial displays. | 1hour
  Emotional facial displays perception measured with a standardized emotional program in terms of congruency (total score and standard deviation).

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Gatignol, Principal Investigator — Laboratoire de physiopathologie respiratoire, UMR_S 1158 INSERM/UPMC " Neurophysiologie Respiratoire Expérimentale et Clinique "
Locations (1):
- Laboratoire de Physiopathologie Respiratoire du Service de Pneumologie et de Réanimation, Paris, France

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT03619720/Prot_SAP_000.pdf